CLINICAL TRIAL: NCT05222750
Title: Epidemiology of Thrombotic Thrombocytopenia Syndrome in Integrated Health-care Database in England.Secondary Data Analysis Using a Cohort Design
Brief Title: Epidemiology of Thrombotic Thrombocytopenia Syndrome in Integrated Health-care Database in England
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8111R00011
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (3):
- Pre-COVID-19
  Interventions: Other: Pre-COVID-19
- COVID-19
  Interventions: Other: COVID-19
- COVID-19 vaccination roll - out
  Interventions: Other: COVID-19 vaccination roll-out

INTERVENTIONS:
Other: Pre-COVID-19 — Pre-COVID-19
  Groups: Pre-COVID-19
Other: COVID-19 — COVID-19
  Groups: COVID-19
Other: COVID-19 vaccination roll-out — COVID-19 vaccination roll-out
  Groups: COVID-19 vaccination roll - out

SUMMARY:
Background/Rationale: A rare syndrome of thrombosis associated with low platelets has been reported in a few cases of recent exposure to COVID-19 vaccine. Medicines & Healthcare products Regulatory Agency (MHRA) had requested for all cases of thrombosis or thrombocytopenia occurring within 28 days of coronavirus vaccine to be reported via the online yellow card system. This syndrome seems to be affecting patients of all ages and both genders; at present there is no clear signal of risk factors. Up to and including 14 April 2021, the MHRA had received 168 United Kingdom (UK) reports of thrombo-embolic events with concurrent low levels of platelets following the use of the COVID-19 Vaccine AstraZeneca. The United Kingdom (UK) is uniquely placed to study this area because of its registration-based primary care system, and a unique identifier number links primary care to secondary care data. Additionally, vaccination is well advanced, maximising population wide vaccine exposure.

Objectives and Hypotheses: Estimate event rates and describe characteristics of patients with a record for thrombotic thrombocytopenia syndrome, thromboembolism or thrombocytopenia, in the general population of England.

Methods:

Study design: Secondary data analysis using a cohort design. Data Source(s): This is a retrospective cohort study using linked secondary databases in England accessed through the NHS Digital Trusted Research Environment (TRE). The primary care data will be linked with vaccination, primary care data, hospitalization, COVID-19 test results, mortality data at the national level for capture of key study variables. This integrated digital health system will also include other linkages such as the Oxford-Royal College of General Practitioners sentinel network; ORCHID.

Study Population: All patients, with our population of interest in England who are present in the integrated health records of NHS Digital TRE and/or the Oxford Royal College of General Practitioners Clinical Informatics Digital Hub (ORCHID) database at the start of each study period.

Variables: Demographic, socioeconomic, clinical descriptors and risk factors for thrombosis and/or thrombocytopenia; COVID-19 vaccines.

Statistical Analysis: The event rates with 95% CIs will be calculated by dividing the number of events with person-time at risk per 100,000 person-years. Further, event count and event rates will be evaluated in a relationship with COVID-19 vaccination date.

ELIGIBILITY:
Inclusion Criteria:

* All patients, with a primary focus from age 16 years old and older, in England who are present in the integrated database at the start of each study period.

Exclusion Criteria:

* Less than 12 months of prior history at start of each respective study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients, with a primary focus from age 16 years old and older, in England who are present in the integrated database at the start of each study period.
Sampling Method: Non-Probability Sample
Enrollment: 41200246 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Estimate event rates and describe characteristics of patients with a record for thrombotic thrombocytopenia syndrome, thromboembolism or thrombocytopenia, in the general population of England. | 9 months
  This is to complete studies in NHS Digital and ORCHID data

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis _Redacted (002).pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111R00011&attachmentIdentifier=6504f229-1baf-4c09-8797-30d6de329073&fileName=Epi_of_TTS_CSR_Synopsis__Redacted_(002).pdf&versionIdentifier=